CLINICAL TRIAL: NCT07187232
Title: Effects of Acupressure on Physiological Indicators, Oxygen Demand and Length of Hospital Stay in Premature Infants With Pulmonary Infiltration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 221235
Record Dates: First submitted 2025-06-26; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: PreTerm Neonate; Pulmonary Complications
Keywords: Acupressure; Preterm Infants; Pulmonary Infiltration; Suction Frequency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure (Experimental)
  Interventions: Behavioral: massage acupoints
- Routine care (Placebo Comparator)
  Interventions: Behavioral: Routine care

INTERVENTIONS:
Behavioral: massage acupoints — The massage acupoints involved Zusanli (ST36), Fenglong (ST40), Zhongfu (LU1), Tanzhong (CV17), and Feishu (BL13). Each acupoint was massaged for 2 minutes, totaling 10 minutes per session. The routine care included chest physiotherapy and sputum suction as needed every 3 hours (PRN, Q3H).
  Arms: Acupressure
Behavioral: Routine care — The routine care included chest physiotherapy and sputum suction as needed every 3 hours (PRN, Q3H).
  Arms: Routine care

SUMMARY:
In 2020, 11.6% of newborns are delivered prematurely in Taiwan. Excessive sputum is a common symptom of respiratory complications in premature infants. Effective methods for reducing sputum secretion in premature infants need to be urgently explored.

ELIGIBILITY:
Inclusion Criteria:

* Newborn ≤32 weeks of gestational age
* X-ray reporting pulmonary infiltration requiring suctioning
* Treated with O2 nasal cannula or High-flow nasal cannula

Exclusion Criteria:

* Congenital pulmonary structural abnormalities
* Muscular weakness
* Heart disease, excluding Patent Ductus Arteriosus(PDA) and Atrial Septal Defect (ASD)
* Abnormal bleeding conditions
* Chest tube placement
* Compromised skin integrity at the acupressure sites

Min Age: 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-07-02 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Frequency of sputum suction | The study outcomes were evaluated before and day 5, day 10, day 12 after the intervention.
  Suctioning frequency per day was obtained from nursing records throughout the intervention period and for the subsequent two days.

SECONDARY OUTCOMES:
Physiological indicatores | These outcomes were recorded 2 days before the intervention, days 1-5 of the intervention, days 6-10 of the intervention, and 2 days after the intervention.
  Physiological indicators include heart rate、 respiratory rate、 oxygen saturation.
  Physiological indicators per day was obtained from nursing records throughout the intervention period and for the subsequent two days on physiological chart record sheets.
  1. Heart Rate Description: Daily heart rate obtained from nursing records. Unit of measure: beats per minute (bpm). Measured instruments: Philips MX450 ECG Monitor.
  2. Respiratory Rate Description: Daily respiratory rate obtained from nursing records. Unit of measure: breaths per minute. Measured instruments: Philips MX450 ECG Monitor.
  3. Oxygen Saturation (SpO₂) Description: Daily oxygen saturation obtained from nursing records. Unit of measure: percentage (%). Measured instruments: Philips MX450 ECG Monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- Taiwan, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No